CLINICAL TRIAL: NCT00997451
Title: Fatigue Self- Management in Primary Care: Efficacy, Credibility, and Economics
Brief Title: Fatigue Self-Management in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIH 5R01NR010229 - 03
Record Dates: First submitted 2009-03-28; First posted 2009-10-19 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Medically Unexplained Chronic Fatigue; Chronic Fatigue Syndrome
Keywords: Medically unexplained chronic fatigue; Chronic fatigue syndrome; Cognitive-behavior therapy; Self-management; Primary care; Nurses; Economic analysis; Cost effectiveness; One year follow-up
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Behavioral Self-Management (Experimental): Cognitive-behavioral self-management
  Interventions: Behavioral: Cognitive-behavioral self-management
- Symptom Monitoring (Active Comparator)
  Interventions: Behavioral: Symptom monitoring
- Standard Medical Care (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive-behavioral self-management — Graded activity, pacing, stress reduction, low effort pleasant activities, cognitive coping skills.
  Arms: Behavioral Self-Management
Behavioral: Symptom monitoring — Daily symptom via web diary
  Arms: Symptom Monitoring

SUMMARY:
This study will evaluate, in a primary care setting, the effectiveness of a brief self-management behavioral treatment in patients with medically unexplained chronic fatigue. The hypothesis will be tested that fatigue self-management will yield improvements in fatigue,functioning, and distress in comparison to the two control conditions: standard medical care alone or standard medical care plus an attention control symptom monitoring condition.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of unexplained chronic fatigue
* diagnosis of chronic fatigue syndrome

Exclusion Criteria:

* medically explained fatigue
* any psychosis or dementia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2009-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scale | 3 months, 6 months, 15 months

SECONDARY OUTCOMES:
Beck Anxiety Inventory | 3 months, 6 months, 15 months
Beck Depression Inventory | 3 months, 6 months, 15 months
SF-36 physical function subscale | 3 months, 6 months, 15 months
Global Impression of Change Rating | 3 months, 6 months, 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Fred Friedberg, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

REFERENCES:
- [Derived] Meng H, Friedberg F, Castora-Binkley M. Cost-effectiveness of chronic fatigue self-management versus usual care: a pilot randomized controlled trial. BMC Fam Pract. 2014 Nov 25;15:184. doi: 10.1186/s12875-014-0184-7. PMID 25421363
- [Derived] Friedberg F, Napoli A, Coronel J, Adamowicz J, Seva V, Caikauskaite I, Ngan MC, Chang J, Meng H. Chronic fatigue self-management in primary care: a randomized trial. Psychosom Med. 2013 Sep;75(7):650-7. doi: 10.1097/PSY.0b013e31829dbed4. Epub 2013 Aug 6. PMID 23922399